CLINICAL TRIAL: NCT01854242
Title: Glycogen Storage Disease Type Ia and Inflammatory Bowel Disease: A New Comorbidity or Secondary Consequence
Brief Title: Study of the Relationship Between Glycogen Storage Disease Type Ia and Inflammatory Bowel Disease
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: Prometheus Laboratories (Industry)
Responsible Party: Sponsor
Other Study IDs: IRB201300312; COL13IBD01 (Other Grant/Funding Number: Prometheus Laboratories/COL13IBD01)
Record Dates: First submitted 2013-05-10; First posted 2013-05-15 (Estimated); Results first posted 2014-12-18 (Estimated); Last update posted 2020-07-28 (Actual); Status verified 2019-02

CONDITIONS: Inflammatory Bowel Disease; Glycogen Storage Disease Type Ia
MeSH Terms: conditions — Inflammatory Bowel Diseases; Hepatorenal form of glycogen storage disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Glycogen Storage Disease type Ia patients: The participants will have one blood draw for this study. The test will be performed on the blood.
  Interventions: Other: Glycogen Storage Disease type Ia patients

INTERVENTIONS:
Other: Glycogen Storage Disease type Ia patients — The participants will have one blood draw for this study. The test will be performed on the blood.
  Other Names: GSD Type Ia

SUMMARY:
The purpose of this research study is to understand the relationship between inflammatory bowel disease (IBD) and Glycogen storage disease (GSD)type Ia. GSD type Ib has been established to have an association with IBD with clinical and histologic features that mirror those of Crohn disease. Development of the disease seems to be related to the defect of neutrophil function in individuals with GSD type Ib and subsequent colonic inflammation. In the last decade, it has become a standard for patients with GSD type Ib and gastrointestinal symptoms to be evaluated for IBD. Patients with GSD type Ia were not recognized to have similar gastrointestinal symptoms until recently. The prevalence of IBD is greater in patients with GSD type Ia versus the general population.

DETAILED DESCRIPTION:
The purpose of this research study is to understand the relationship between IBD and GSD type Ia. The Investigators will be attempting to develop a blood test which will be aimed at the participants diagnosis of IBD.

As a participant in this research study, a blood sample will be collected during your admission to the University of Florida. This will not affect the length of stay of your scheduled visit. There will be no scheduled clinic follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Anyone with Glycogen Storage Disease type Ia

Exclusion Criteria:

* Anyone where the amount of blood needed to complete the Prometheus test exceeds 3ml/kg.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Glycogen storage disease (GSD) type I is an autosomal recessive disorder of glycogen metabolism that affects approximately 1 in 100,000 live births (1). Mutations of the genes that encode glucose 6-phosphatase [type Ia] (2) and glucose 6-phosphate translocase [type Ib] (3) have been isolated. Diagnosis is usually suspected in infants with fasting hypoglycemia, lactic acidosis, hyperlipidemia, and hepatomegaly. Other features include stomatitis, growth retardation, osteopenia and hyperuricemia.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2013-11; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicole T Lawrence, MD, Principal Investigator — University of Florida; David A Weinstein, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida and Shands, Gainesville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Glycogen Storage Disease Type Ia Patients
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Glycogen Storage Disease Type Ia Patients
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 32
  Between 18 and 65 years | 18
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 27
Region of Enrollment [Number; unit: participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Serologic, Genetic and Inflammatory Markers Consistent With Inflammatory Bowel Disease
Description: Participants who tested positive for Crohn disease, ulcerative colitis, or unspecified inflammatory bowel disease (IBD) on a panel for IBD are reported in the Outcome Measure Data Table.
Time Frame: 2 weeks
Measure: Number; unit: participants testing positive
Arm/Group | Glycogen Storage Disease Type Ia Patients
Number analyzed (Participants) | 50
participants testing positive | 11

ADVERSE EVENTS:
Arm/Group | Glycogen Storage Disease Type Ia Patients
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No